CLINICAL TRIAL: NCT01852032
Title: Computed Tomography Versus Standard 2D Mammography Versus 3D Tomosynthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 221183
Record Dates: First submitted 2012-10-29; First posted 2013-05-13 (Estimated); Results first posted 2018-03-16 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Breast cancer Patients (Experimental): Tomosynthesis Breast Scanning is done and breast CT Scanning is done.
  Interventions: Radiation: Tomosynthesis Breast Scanning; Radiation: Breast CT Scanning

INTERVENTIONS:
Radiation: Tomosynthesis Breast Scanning — The breast is positioned and compressed the same way it is in a conventional mammogram using a compression paddle device. The subject will be instructed to hold their breath and not move during the 7- second 3-D tomosynthesis acquisition. The affected breast is positioned with MLO compression. The radiation dose levels for each scan are equivalent to mammography
Radiation: Breast CT Scanning — CT scanning will be performed before and after I.V. iodine contrast injection. The subject will lie prone on a large table (which is covered by a foam pad), and she will place the breast to be scanned in a small hole in that tabletop. The hole is surrounded by a soft neoprene "hammock," which will allow the subject's entire upper torso to slump into the scan plane of the device. After positioning of the affected breast by a female mammography technologist, the subject will be instructed to hold their breath for 16 seconds and the pre-contrast scan will commence. There will be no breast compression. Other than the sound of the relatively noisy x-ray system in the room, the subject will not feel or sense any aspect of this scan.

SUMMARY:
The purpose of this study is to compare the imaging performance of an investigational breast computed tomography (CT) scanner, built at UC Davis, with that of an FDA-Approved breast tomosynthesis scanner (capable of producing standard 2-D mammography and 3-D tomosynthesis images), built by Hologic, Incorporated, in a group of patients with suspected breast cancer.

DETAILED DESCRIPTION:
The primary aim of this study is the comparison of Beta values of several different CT and Tomosynthesis views (Beta of CT Sagittal View, Beta of CT Coronal View, Beta of CT Axial View, Beta of Tomosynthesis Craniocaudal View, Beta of Tomosynthesis Medial Lateral Oblique View). Lower Beta values correspond to better image quality (less noise, increased cancer detection).

ELIGIBILITY:
Inclusion Criteria:

* 35 years of age or older
* While male patients will not be explicitly excluded, it is expected that all patients in this study will be women
* Diagnostic findings from prior mammography suspicious for, or highly suggestive of, breast malignancy -BIRADS (Breast Imaging Reporting and Data System) categories 4 and 5
* Scheduled for ultrasound or stereotactic core biopsy
* Ability to lie still on a table top for up to 10 minutes, longer than the typical breast CT duration.
* Ability to understand risks, procedures, and benefits involved

Exclusion Criteria:

* Recent breast biopsy
* History of breast augmentation implant
* Pregnant or Positive urine pregnancy test (UPT) or currently breast-feeding
* History of moderate or severe adverse reaction to iodinated contrast injection
* Recent serum creatinine ≥ 1.5 mg/dL
* History of Diabetes Mellitus
* Currently taking Glucophage or Glucovance (Metformin)
* History of chronic asthma
* History of allergy to iodine
* Multiple food and/or drug allergy
* Renal disease
* History of pulmonary disease, phobia of breath holding, or other condition that could prevent the subject from being able to perform the 16 second breath hold

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-11; Primary Completion 2016-03-04 (Actual); Study Completion 2016-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M Boone, PhD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Breast Cancer Patients
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Female participants over the age of 35 with suspected breast cancer
Arm/Group | Breast Cancer Patients
Number analyzed (Participants) | 23
Age, Customized [Number; unit: participants]
  greater than 35 years old | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Beta of CT Coronal View
Description: frequency range corresponding to noise power spectrum (NPS) where beta = NPS(f) = af^-B.
  beta is calculated as noise corresponding to frequency. The values of the exponent, beta, range from 1.5 to 3.5 Lower Beta values correspond to better image quality (less noise, increased cancer detection).
Time Frame: Day 1
Population: Participants with suspected breast cancer
Measure: Mean (Standard Deviation); unit: power-law slope(B)
Arm/Group | Breast Cancer Patients
Number analyzed (Participants) | 23
power-law slope(B) | 1.75 (0.424)

2. Primary Outcome: Beta of CT Sagittal View
Description: as for outcome 1
Time Frame: Day 1
Population: Participants with suspected breast cancer
Measure: Mean (Standard Deviation); unit: power-law slope(B)
Arm/Group | Breast Cancer Patients
Number analyzed (Participants) | 23
power-law slope(B) | 1.83 (0.352)

3. Primary Outcome: Beta of CT Axial View
Description: as for outcome 1
Time Frame: Day 1
Population: Participants with suspected breast cancer
Measure: Mean (Standard Deviation); unit: power-law slope(B)
Arm/Group | Breast Cancer Patients
Number analyzed (Participants) | 23
power-law slope(B) | 1.79 (0.397)

4. Primary Outcome: Beta of Tomosynthesis Craniocaudal View
Description: as for outcome 1
Time Frame: Day 1
Population: Participants with suspected breast cancer
Measure: Mean (Standard Deviation); unit: power-law slope(B)
Arm/Group | Breast Cancer Patients
Number analyzed (Participants) | 23
power-law slope(B) | 3.06 (0.361)

5. Primary Outcome: Beta of Tomosynthesis Medial Lateral Oblique View
Description: as for outcome 1
Time Frame: Day 1
Population: Participants with suspected breast cancer
Measure: Mean (Standard Deviation); unit: power-law slope(B)
Arm/Group | Breast Cancer Patients
Number analyzed (Participants) | 23
power-law slope(B) | 3.10 (0.315)

ADVERSE EVENTS:
Arm/Group | Breast Cancer Patients
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No